CLINICAL TRIAL: NCT06179238
Title: Education Given to Patients With Urinary Catheters on Urinary Catheter Self-care Management and Urinary Tract Infection Impact on Status
Brief Title: Urinary Catheter Self-care Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Filz Ozel Cakir, Assistant professor, Kastamonu University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12345
Record Dates: First submitted 2023-11-19; First posted 2023-12-21 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Chronic Diseases
MeSH Terms: conditions — Chronic Disease | interventions — Educational Status; Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with urinary catheter receiving patient education (Other): The population of the study consisted of urinary catheterized patients treated in the clinics of a Training and Research Hospital. G*Power power analysis was used to calculate the number of individuals constituting the sample. The effect size was set to 0.80, which is a high level according to Cohen for comparing the means of independent samples. To ensure that the statistical power of the study was above 95%, the sample size was set at a 5% significance level and the effect size was 0.5. (df = 68; t = 1.668) The sample size was calculated as 70 patients. The study is planned to be conducted with 35 patients for each of the two study groups.
  Interventions: Other: Education
- Patient with urinary catheter without patient education (Other): The population of the study consisted of urinary catheterized patients treated in the clinics of a Training and Research Hospital. G*Power power analysis was used to calculate the number of individuals constituting the sample. The effect size was set to 0.80, which is a high level according to Cohen for comparing the means of independent samples. To ensure that the statistical power of the study was above 95%, the sample size was set at a 5% significance level and the effect size was 0.5. (df = 68; t = 1.668) The sample size was calculated as 70 patients. The study is planned to be conducted with 35 patients for each of the two study groups.
  Interventions: Other: without patient education

INTERVENTIONS:
Other: Education — Patients with urinary catheter insertion during the study periods will be identified and consent will be obtained for the study. In the first stage of the study, questionnaires will be applied face to face to the experimental group and the control group. Then, education and brochures will be given to the patients in the experimental group. Patients in the experimental group will be visited and evaluated every day until the urinary catheter is removed. After the urinary catheter is removed, the patients in the experimental group and urinary catheter self-care management scale will be applied to the control group.
  Arms: Patient with urinary catheter receiving patient education
Other: without patient education — without patient education
  Arms: Patient with urinary catheter without patient education

SUMMARY:
It is important for healthcare professionals to be sensitive to the needs of patients undergoing urinary catheterization. Patients and their relatives should be educated, guided and supported by nurses and other healthcare professionals. The aim of this study was to determine the effect of education given to patients with urinary catheterization on urinary catheter self-care management and urinary tract infection status. is planned as an experimental research.

DETAILED DESCRIPTION:
The most important risk factor in the development of healthcare-associated infections of the urinary system is the insertion of a urinary catheter. Because when a urinary catheter is inserted, the possibility of developing daily bacteriuria inthe patient increases. Urinary catheter application can cause the development of fungal infections as well as bacterial infections in the patient. Although most of these infections are asymptomatic and do not pose a threat, symptomatic serious infections rarely occur. may occur. There is a risk of catheter-associated urinary tract infection in both long and short-term catheterization. This risk increases as the duration of catheterization increases. According to the Nursing Regulation published in 2011 in our country, the initiatives in this direction are expected to be continued by nurses. Therefore, in this study, the knowledge and practices of patients with urinary catheter will be examined and the effect of the education given on urinary catheter self-care management and urinary tract infection status will be evaluated. It is thought that the results of the study will guide patients with urinary catheters and nurses who provide care about the care and education of patients.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* Urinary catheterization
* Being conscious
* To be able to do self-care

Exclusion Criteria:

* Not volunteering to participate in the study
* Lack of awareness
* Inability to take care of themselves

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
The Urinary Catheter Self-Care Management Scale | 10 days
  The Urinary Catheter Self-Care Management Scale consists of a total of 13 items and 4 sub-dimensions.Urinary Catheter Self-Efficacy was funded by the United States National Institute of Nursing Research and developed by Wilde et al. in 2016. The scale consists of a total of 13 items and 4 subscales. The sub-dimensions of the scale are related to physician/nurse communication (items: items 7, 8, 9 and 13), avoid restriction of daily activities (items 10, 11 and 12), prevention of catheter dislodgement (items 4, 5 and 6) and self-efficacy/ fluid intake (items 1, 2 and 3). Scale items are scored on a 10-point Likert scale ranging from 1 = "I am not at all sure that I can do it" to 10 = "I am not at all sure that I can do it". "I am completely sure that I can do it" and high scores indicate high self-efficacy. is a good measure of the quality of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu Training and Research Hospital, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided